CLINICAL TRIAL: NCT02342782
Title: Phase I Study of Yttrium-90 Labeled Anti-CD25 Monoclonal Antibody Plus Standard BEAM Conditioning for Autologous Hematopoietic Cell Transplantation in Patients With Mature T-Cell Non-Hodgkin Lymphoma: the aTAC BEAM Regimen
Brief Title: Yttrium Y 90 Basiliximab and Combination Chemotherapy Before Stem Cell Transplant in Treating Patients With Mature T-cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14349; NCI-2015-00019 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14349 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Recurrent Mature T- and NK-Cell Non-Hodgkin Lymphoma; Refractory Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Recurrent Cutaneous T-Cell Non-Hodgkin Lymphoma; Refractory Cutaneous T-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, T-Cell, Cutaneous | interventions — Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (yttrium Y 90 basiliximab, BEAM, AHCT) (Experimental): Patients receive yttrium Y 90 basiliximab IV on days -21 and -14, carmustine IV over 1-2 hours on days -7 and -6, cytarabine IV BID on days -5 to -2, etoposide IV BID on days -5 to -2, and melphalan IV on day -1. Patients undergo autologous hematopoietic stem cell transplant on day 0.
  Interventions: Biological: Yttrium Y 90 Basiliximab; Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Biological: Yttrium Y 90 Basiliximab — Given IV
  Other Names: 90Y Basiliximab
Drug: Carmustine — Given IV
  Other Names: FDA 0345; BCNU; BiCNU
Drug: Etoposide — Given IV
  Other Names: Lastet; VP-16
Drug: Cytarabine — Given IV
  Other Names: CHX-3311; U-19920; Ara-C; Cytosar
Drug: Melphalan — Given IV
  Other Names: Alkeran; L-PAM
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo AHCT
  Other Names: Autologous Stem Cell Transplantation
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of yttrium Y 90 basiliximab when given together with standard combination chemotherapy before a stem cell transplant in treating patients with mature T-cell non-Hodgkin lymphoma. Radioactive substances linked to monoclonal antibodies, such as yttrium Y 90 basiliximab, can bind to cancer cells and give off radiation which may help kill cancer cells. Drugs used in chemotherapy, such as carmustine, cytarabine, etoposide, and melphalan (BEAM), work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving yttrium Y 90 basiliximab and chemotherapy before a stem cell transplant may help kill any cancer cells that are in the body and help make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. Stem cells that were collected from the patient's blood and stored before treatment are later returned to the patient to replace the blood-forming cells that were destroyed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if administration of 90Y-basiliximab/DOTA (yttrium Y 90 basiliximab), when given in combination with standard dose BEAM, as conditioning for autologous hematopoietic cell transplant (AHCT), is safe, by evaluation of toxicities, including type, frequency, severity, attribution, time course and duration.

II. To determine the maximum tolerated dose (MTD) of 90Y-basiliximab/DOTA when given in combination with standard dose BEAM, in patients with T-cell non-Hodgkin lymphoma (T-NHL) as part of conditioning for AHCT.

SECONDARY OBJECTIVES:

I. To characterize and evaluate hematologic recovery in terms of neutrophil and platelet engraftment time.

II. To estimate radiation doses to the whole body and normal organs through serial imaging studies.

III. To estimate overall survival, progression-free survival, non-relapse mortality and cumulative incidence of relapse/progression at 100-days (non-relapse mortality [NRM] only), 1-year and 2-years.

OUTLINE: This is a dose-escalation study of yttrium Y 90 basiliximab.

Patients receive yttrium Y 90 basiliximab intravenously (IV) on days -21 and -14, carmustine IV over 1-2 hours on days -7 and -6, cytarabine IV twice daily (BID) on days -5 to -2, etoposide IV BID on days -5 to -2, and melphalan IV on day -1. Patients undergo autologous hematopoietic stem cell transplant on day 0.

After completion of study treatment, patients are followed up at 30, 100, and 180 days and 1, 1.5, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pathologically confirmed diagnosis of systemic mature T-cell non-Hodgkin lymphoma (NHL) with City of Hope pathology review as per World Health Organization (WHO) classification of lymphomas 2008, who are deemed eligible for high dose therapy and AHCT including patients in:

  * T-NHL histologies including peripheral T-cell lymphomas (PTCLs), cutaneous T-cell lymphomas (CTCLs) and natural killer (NK)/T cell lymphomas
  * First remission after initial first-line therapy (CR1) in PTCL patients, except for anaplastic lymphoma receptor tyrosine kinase (ALK)+ anaplastic large cell lymphoma (ALCL) and CTCL; patients with minimal residual disease after induction therapy may also be eligible at the discretion of the principal investigator (PI)
  * Relapsed/refractory disease, stable disease, partial remission (PR) or complete remission (CR), who have received at least 2 lines of therapy, and do not have an adequate allogenetic stem cell transplant option
* Life expectancy >= 6 months
* Karnofsky status >= 70%
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Cardiac ejection fraction of >= 50% by echocardiogram or multi gated acquisition scan (MUGA)
* Forced expiratory volume in one second (FEV1) > 65% of predicted measured, or diffusing capacity of the lung for carbon monoxide (DLCO) > 50% of predicted measured
* Bilirubin < 1.5 x normal except in cases where abnormal liver function tests (LFTS) are due to involvement with T-NHL
* Serum glutamic oxaloacetic transaminase (SGOT) AND serum glutamate pyruvate transaminase (SGPT) < 2 x normal except in cases where abnormal LFTS are due to involvement with T-NHL
* Serum creatinine of < 1.5 mg/dL, and a measured creatinine clearance of > 60 mL/min
* Patients will be enrolled at collection of at least 3.0 x 10^6 CD34 cells/kg of autologous hematopoietic progenitor cells (HPC-A) by apheresis; a minimum of 2 collection procedures is required, unless collection on day # 1 > 5.0 x 10^6, CD34 cells/kg; a maximum of 10 collections is allowed; bone marrow harvest to supplement apheresis is not allowed
* Recovery from non-hematologic toxicities of salvage cytoreductive chemotherapy to =< grade 2 (Common Terminology Criteria for Adverse Events [CTCAE] version 4 [v4])
* Body mass index (BMI) > 35% will be considered on a case-by-case basis by the Radiation Oncology principal investigator (P.I.)
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Systemic chemotherapy or radiation cannot have been given within 4 weeks prior to the Y-90 dose of radioimmunotherapy (RIT), with the exception of single agent cyclophosphamide priming chemotherapy administered for mobilization

Exclusion Criteria:

* Progressive disease
* Patients should not have any uncontrolled illness including ongoing or active infection requiring therapy
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy; may have received an experimental agent prior to enrolling in the trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to basiliximab
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with indium In 111 (111In-) and 90Y-basiliximab-DOTA
* Prior high dose chemotherapy for autologous hematopoietic cell transplantation or prior allogeneic transplantation
* Significant prior external beam dose-limiting radiation to a critical organ based on review of the prior radiation treatment records by the Radiation Oncology PI; patients who have had prior external beam radiation > 2000 cGy (at 180 to 200 cGy per day) to the lung will be ineligible; patients with ANY prior radiation to the heart are ineligible; patients with > 500 cGy to the kidney will be excluded from the study; Note: patients who have had electron beam therapy are still eligible and will be evaluated on a case by case basis by the Radiation Oncology PI
* Presence of antibody against basiliximab in serum (only required for patients who have received prior antibody)
* Research participants with presence of other active malignancy; however, research participants with history of prior malignancy treated with curative intent and in complete remission are eligible; any history of myelodysplasia is excluded
* Active hepatitis B or C viral infection or hepatitis B surface antigen positive
* Patients with a detectable human immunodeficiency virus (HIV) viral load or who are HIV-positive AND have a resistant genotype
* Patients with psychosocial circumstances or illnesses that preclude protocol participation (to be determined by P.I.)
* Any cytogenetic abnormality in the bone marrow that is known to be associated with or predictive of myelodysplasia is excluded; this includes, but is not limited to, del(5), del(7), del(11)
* Evidence of marrow disease by flow and morphology after upfront or salvage cytoreductive therapy and before stem cell mobilization
* Bone marrow (BM) harvest required to reach adequate cell dose for transplant
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
MTD of yttrium Y 90 basiliximab defined as the highest dose in which fewer than 33% of patients experience dose limiting toxicity attributable to study treatment, among those evaluable for toxicity | 30 days post-transplant
  Dose limiting toxicities will be graded by the Modified Bearman scale.
Incidence of toxicities assessed using National Cancer Institute (NCI) CTCAE version 4.03 | Up to 100 days post-transplant
  Observed toxicities will be summarized by type (organ affected or laboratory determination such as absolute neutrophil count), severity (by NCI CTCAE version 4.03 and nadir or maximum values for lab measures), date of onset, duration, reversibility, and attribution.

SECONDARY OUTCOMES:
Disease response by Cheson 2007 criteria | Up to 2 years post-transplant
Engraftment: neutrophil and platelet recovery | Up to 2 years post-transplant
Overall survival | From start of therapy (stem cell infusion) to death from any cause, assessed up to 2 years post-transplant
  Survival estimates will be calculated using the Kaplan-Meier method.
Progression-free survival | From start of therapy (stem cell infusion) to the first observation of disease relapse/progression or death from any cause, assessed up to 2 years post-transplant
  Survival estimates will be calculated using the Kaplan-Meier method.
Non-relapse mortality | From start of therapy until non-disease related death, or last follow-up, whichever comes first, assessed up to 2 years post-transplant
  The cumulative incidence of relapse/progression and non-relapse mortality will be calculated as competing risks using the Gray method.
Cumulative incidence of relapse/progression | From start of therapy (stem cell infusion) to the first observation of disease relapse/progression, assessed up to 2 years post-transplant
  The cumulative incidence of relapse/progression and non-relapse mortality will be calculated as competing risks using the Gray method.
Absorbed radiation dose to organs assessed by nuclear scan images | Up to day -14

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Zain, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Zain J, Tsai NC, Palmer J, Simpson J, Adhikarla V, Bading JR, Yazaki P, Smith EP, Dandapani S, Song JY, Karras NA, Herrera AF, Salhotra A, Nademanee AP, Nakamura R, Smith DL, Yamauchi D, Poku EK, Biglang-Awa VE, Colcher D, Shively JE, Wu AM, Forman SJ, Wong J, Thomas S. Yttrium-90 anti-CD25 BEAM conditioning for autologous hematopoietic cell transplantation in Peripheral T-cell lymphoma. Blood Adv. 2024 Sep 24;8(18):4812-4822. doi: 10.1182/bloodadvances.2023012497. PMID 38838232